CLINICAL TRIAL: NCT04972916
Title: Patient Navigation-based Tobacco Harm Reduction Program Among Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Tongyao Fan, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00017696
Record Dates: First submitted 2021-06-29; First posted 2021-07-22 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Tobacco Use
Keywords: cancer patients; tobacco harm reduction; patient navigation
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Navigation-based Tobacco Harm Reduction Intervention (Other): All participants will receive a smoking cessation educational brochure and patient navigation intervention delivered over 2 months.
  Interventions: Other: Patient navigation-based tobacco harm reduction intervention

INTERVENTIONS:
Other: Patient navigation-based tobacco harm reduction intervention — At the first intervention interview, the patient navigators will educate participants about the benefits of quitting, introduce smoking cessation resources, motivate participants to link with treatment, help participants attend smoking cessation treatments, and assess barriers that prevented them from being able to consider smoking cessation. The cessation treatment resources will be discussed include PennState Health Smoking Cessation Clinic, Pennsylvania Quitline, or visiting their primary care provider (PCP) to discuss cessation, prescription medications, and/or nicotine replacement therapy. A follow-up call will be made 1 month later to further assist and motivate to use tobacco treatment services, and assess interim tobacco treatment engagement outcome.

SUMMARY:
The purpose of this study is to examine the feasibility and preliminary efficacy of patient navigation to promote linkage to smoking cessation treatments in cancer patients.

DETAILED DESCRIPTION:
The investigators plan to conduct a 2-month 1-arm intervention study that will recruit up to 20 smoking cancer patients at Penn State Cancer Institute. All participants will receive a smoking cessation educational brochure and patient navigation intervention (in-person or by phone) delivered over two months. At the first intervention interview, the patient navigators will educate participants about the benefits of quitting, introduce smoking cessation resources, motivate participants to link with treatment, help participants attend smoking cessation treatments, and assess barriers that prevented them from being able to consider smoking cessation. The cessation treatment resources will be discussed include PennState Health Smoking Cessation Clinic, Pennsylvania Quitline, or visiting their primary care provider (PCP) to discuss cessation, prescription medications, and/or nicotine replacement therapy. A follow-up call will be made 1 month later to further assist and motivate to use tobacco treatment services, and assess interim tobacco treatment engagement outcome. At 2 months after baseline, the final questionnaire will be administered to assess participants' smoking behaviors, engagement in tobacco treatments, and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years of age
* Diagnosis of cancer
* Current cigarette smoker (smoked cigarettes in last 30 days)
* Be able to read and speak English

Exclusion Criteria:

* Age: < 18 years of age
* Unable to read and speak English
* Actively using evidence-based smoking cessation treatments
* Known decisional impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Participant recruitment efficiency and retention rate | From baseline to completion of final assessment, approximately 2 months
  This outcome is measured by the ability to recruit and enroll 20 participants for the 2-month program, individual participant attendance in patient navigation intervention visits, and completion of final assessment.
Acceptability of intervention will be measured by likert-scale questions assessing helpfulness and satisfaction with intervention sessions, feedback on the intervention sessions, and smoking perceptions and behaviors changes | At the final assessment, 2 months after baseline. The changes in smoking perceptions and behaviors will be compared between baseline and final assessments.
  Acceptability will be measured by Likert-scale questions assessing helpfulness and satisfaction with patient navigation intervention sessions, feedback on the intervention sessions, and smoking perceptions and behaviors changes including perceptions of risk, nicotine dependence, stage of change.

SECONDARY OUTCOMES:
Number of participants engaged in tobacco treatments | At the final assessment, 2 months after baseline
  Engagement is defined as completion at least one tobacco cessation counseling session OR use of at least one FDA-approved cessation medication for at least 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: Tongyao Investigator, MPH, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided